CLINICAL TRIAL: NCT00304369
Title: The Response of Clostridium Difficile Infection to Metronidazole Therapy
Brief Title: Response of Clostridium Difficile Infection to Metronidazole Therapy
Status: Completed | Type: Observational
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Daniel M. Musher MD, Principle Investigator, Michael E. DeBakey VA Medical Center
Other Study IDs: H-16175
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Clostridium Enterocolitis; Pseudomembranous Colitis; Antibiotic-Associated Colitis
Keywords: Clostridium difficile
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Metronidazole

SUMMARY:
In this record review study, our objective is to determine the rates of cure, failure and relapse following treatment of C. difficile colitis with metronidazole.

DETAILED DESCRIPTION:
Clostridium difficile is a major cause of nosocomial infection. When this organism proliferates in the colon, usually as a result of prior antibiotic therapy in a hospitalized or otherwise debilitated person, a variety of potentially serious consequences follow, such as fever, leukocytosis, abdominal pain, diarrhea and ileus. Some patients require surgical exploration and colectomy, and our hospital has had several deaths attributable to C. difficile colitis in the past year.

C. difficile colitis is treated with metronidazole, and earlier literature on this subject, written in the 1980's and early 1990s, suggests that the response rate is excellent, exceeding 90-95%. Our clinical observation has suggested that treatment with metronidazole is followed by a surprisingly high rate of failure, perhaps 25-30%. The clinical problem is that there are, at present, no desirable alternatives. Vancomycin, given orally, is said to be highly effective in treating this infection, but this may not be true, and the administration of this drug is associated with emergence of vancomycin-resistant bacteria, a major problem in modern hospitals. No other drug is approved for treatment of C. difficile infection.

We believe it is important to determine the actual rate of failure of treatment with metronidazole. This will provide an impetus for developing new therapeutic approaches.

We will review the records of patients who have been treated for confirmed C. difficile infection with metronidazole at the VAMC for the past 12 months in order to determine the rates of cure, failure, and relapse following therapy. This is a simple record review study to determine if our clinical suspicion is correct, namely, if the rate of failure of metronidazole therapy is much higher than that reported in the medical literature of 10-15 years ago.

ELIGIBILITY:
Inclusion Criteria:

* records of patients who have a fecal sample positive for C. difficile toxin and who are then treated for C. difficile colitis with oral metronidazole will be included in this study.

Exclusion Criteria:

* Patients who did not receive at least 7 days of metronidazole

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. Debakey VA Medical Center, Houston, Texas, United States